CLINICAL TRIAL: NCT02289833
Title: A Phase 2, Multicenter, Single-Arm Study of Trastuzumab Emtansine in Patients With HER2 IHC-Positive, Locally Advanced or Metastatic Non-Small Cell Lung Cancer Who Have Received At Least One Prior Chemotherapy Regimen
Brief Title: A Study of Trastuzumab Emtansine in Participants With Human Epidermal Growth Factor Receptor (HER)2 Immunohistochemistry (IHC)-Positive, Locally Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BO29389; 2014-001237-83 (EudraCT Number)
Record Dates: First submitted 2014-11-04; First posted 2014-11-13 (Estimated); Results first posted 2017-11-22 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-07

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Ado-Trastuzumab Emtansine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort IHC2+ (Experimental): Participants with HER2 IHC2-positive (IHC 2+) locally advanced or metastatic NSCLC, who had received at least one prior platinum-based chemotherapy regimen, will receive trastuzumab emtansine.
  Interventions: Drug: Trastuzumab Emtansine
- Cohort IHC3+ (Experimental): Participants with HER2 IHC3-positive (IHC 3+) locally advanced or metastatic NSCLC, who had received at least one prior platinum-based chemotherapy regimen, will receive trastuzumab emtansine.
  Interventions: Drug: Trastuzumab Emtansine

INTERVENTIONS:
Drug: Trastuzumab Emtansine — Trastuzumab emtansine will be administered intravenously (IV) at a dose of 3.6 mg/kg on Day 1 of every 21-day cycle until disease progression (as assessed by the investigator), unmanageable toxicity, or study termination by the sponsor, whichever occurs first.
  Other Names: Kadcyla, T-DM1

SUMMARY:
This is a Phase 2, multicenter study designed to evaluate the efficacy and safety of trastuzumab emtansine administered as a single-agent in participants with HER2-positive (HER2 IHC 2+ or HER2 IHC 3+) advanced or metastatic NSCLC. Participants will be treated with trastuzumab emtansine administered intravenously at a dose of 3.6 milligrams per kilogram (mg/kg) on Day 1 of 21-day cycles until disease progression (as assessed by the investigator), unmanageable toxicity, or study termination by the Sponsor, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented diagnosis of Stage IIIB not amenable to radical treatment or Stage IV NSCLC (pathological characterization must determine the non-squamous or squamous histological subtype as well as adenocarcinoma subtype classification)
* HER2 status of IHC 2+ or 3+ as determined by a Sponsor-designated central laboratory
* Prior treatment with at least one regimen of platinum-based (cisplatin or carboplatin) chemotherapy in the locally advanced or metastatic setting/recurrent NSCLC with documented disease progression by investigator assessment
* Participants with a known anaplastic lymphoma kinase (ALK) fusion oncogene (must be documented in the participant's chart) must have also experienced disease progression or intolerance with a first-line ALK Tyrosine Kinase Inhibitor (TKI) approved for the treatment of ALK fusion oncogene NSCLC (for example, crizotinib). Disease progression or intolerance must be documented
* Participants with a known mutation in the epidermal growth factor receptor (EGFR) gene (must be documented in the participant's chart) must have also experienced disease progression or intolerance with an EGFR TKI approved for the treatment of EGFR-mutant NSCLC (for example, gefitinib, erlotinib, afatinib). Disease progression or intolerance must be documented
* Measurable disease determined as per the RECIST v1.1
* Life expectancy of at least (>/=) 12 weeks
* Adequate organ function
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Left ventricular ejection fraction (LVEF) >/= 50 percent (%) by either echocardiogram (ECHO) or multiple-gated acquisition (MUGA) scan
* Use of highly effective contraception

Exclusion Criteria:

Cancer-Related Criteria:

* Any approved anti-cancer therapy less than or equal to (</=) 21 days (including chemotherapy or hormonal therapy) before the first study treatment; the following exceptions are allowed: (1) TKIs approved for the treatment of NSCLC must be discontinued greater than (>) 7 days prior to the first study treatment on D1C1 (The baseline computed tomography [CT] scan must be completed after discontinuation of TKIs); (2) Hormone-replacement therapy or oral contraceptives; (3) Anti-emetics, Granulocyte-colony stimulating factor (GCS-F), and prophylactic antibiotics according to local standards
* Investigational therapy participation in another clinical study with therapeutic intent </= 21 days before first study treatment
* Previous irradiation is permitted if >/=14 days since the last fraction of radiotherapy have elapsed before the first study treatment on Day 1 as long as a sufficient number of target lesions remain to allow for measurable disease as per RECIST v1.1
* Participants who have untreated brain metastases or are symptomatic; participants with treated brain metastases must have discontinued corticosteroid therapy and not have any neurological symptoms
* History of intolerance (including Grade 3 or 4 infusion reaction) or hypersensitivity to trastuzumab or murine proteins or any excipient of the product
* History of exposure to the following cumulative doses of anthracyclines: Doxorubicin or liposomal doxorubicin > 500 milligram per meter-square (mg/m^2); Epirubicin > 900 mg/m^2; Mitoxantrone > 120 mg/m^2. If another anthracycline, or more than one anthracycline, has been used, the cumulative dose must not exceed the equivalent of 500 mg/m^2 doxorubicin
* Peripheral neuropathy of Grade >/= 3 per the National Cancer Institute Common Toxicity Criteria for Adverse Events Version 4.0 (NCI CTCAE v. 4.0)
* History of other malignancy within the last 5 years, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, Stage I uterine cancer, or other cancers with a similar outcome as those mentioned above

Cardiopulmonary Function Criteria:

* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures
* Severe dyspnea at rest due to complications of advanced malignancy or requiring current continuous oxygen therapy
* Clinical history of active hemoptysis
* Evidence of active pneumonitis during screening
* Current unstable ventricular arrhythmia requiring treatment
* History of symptomatic congestive heart failure (CHF) New York Heart Association (NYHA) classes II-IV
* History of myocardial infarction or unstable angina within 6 months of enrollment
* History of a decrease in LVEF to <50%

General Criteria:

* Current severe, uncontrolled systemic disease (for example, clinically significant cardiovascular, pulmonary, or metabolic disease)
* Major surgical procedure or significant traumatic injury within 28 days before enrollment or anticipation of the need for major surgery during the course of study treatment
* Current pregnancy or lactation
* Current known active infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2014-12-15 (Actual); Primary Completion 2016-10-25 (Actual); Study Completion 2018-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (23):
- United States (5):
  - Cancer Specialists; North Florida ;Jacksonville (AC Skinner Pkwy), Jacksonville, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Karmanos Cancer Institute, Detroit, Michigan
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Seattle Cancer Care Alliance, Seattle, Washington
- Germany (5):
  - HELIOS Klinikum Emil von Behring Klinik f.Pneumologie Onkologie u.Infektiologie, Berlin
  - Kaiserswerther Diakonie Florence Nightingale-Krankenh. Tagesklinik f.Onkologie, Düsseldorf
  - Asklepios-Fachkliniken Muenchen-Gauting; Onkologie, Gauting
  - Krankenhaus Martha-Maria Halle-Doelau gGmbH; Klinik fuer Innere Medizin II, Halle
  - Fachklinik für Lungenerkrankungen, Immenhausen
- Italy (2):
  - Azienda Ospedaliera Univ Parma; Dept Oncologia Medica, Parma, Emilia-Romagna
  - Istituto Europeo Di Oncologia, Milan, Lombardy
- Poland (3):
  - Medical University of Gdansk, Gdansk
  - Mazowieckie Centrum Leczenia Chorob Pluc I Gruzlicy; Oddzial Iii, Otwock
  - Centrum Onkologii - Instytut im. Marii Skłodowskiej-Curie Klinika Nowotworów Piersi i Chirurgii, Warsaw
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center - Oncology, Seoul
- Spain (4):
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona
  - Hospital Ramon y Cajal; Servicio de Oncologia, Madrid
  - Hospital Universitario La Paz; Servicio de Oncologia, Madrid
  - Hospital Clinico Universitario Lozano Blesa; Servicio de Oncologia, Zaragoza
- Switzerland (2):
  - CHUV; Departement d'Oncologie, Lausanne
  - UniversitätsSpital Zürich; Zentrum für Hämatologie und Onkologie, Klinik für Onkologie, Zurich

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened centrally for HER2 status, using archived tumor specimens from previously collected tissue, if available.
Period: Overall Study
Arm/Group | Cohort IHC2+ | Cohort IHC3+
Started | 29 | 20
Completed | 2 | 3
Not Completed | 27 | 17
Not completed — Study discontinuation | 0 | 1
Not completed — Lost to Follow-up | 4 | 0
Not completed — Death | 23 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort IHC2+ | Cohort IHC3+ | Total
Number analyzed (Participants) | 29 | 20 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (10.3) | 61.4 (8.6) | 62.4 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 7 | 20
  Male | 16 | 13 | 29

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Objective Response as Per Investigator Assessment According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v. 1.1)
Description: Objective response is defined as a complete response (CR) or partial response (PR) determined on two consecutive assessments ≥ 4 weeks apart, based on investigator assessment according to RECIST, Version 1.1. CR: disappearance of all target lesions; and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 millimeters (mm). PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: From Day 1 to disease progression (PD) or death from any cause, up to the clinical cutoff date (approximately 22 months)
Population: The efficacy-evaluable population included participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort IHC2+ | Cohort IHC3+
Number analyzed (Participants) | 29 | 20
percentage of participants | 0 [0 to 11.9] | 20.0 [5.7 to 43.7]

2. Secondary Outcome: Percentage of Participants Who Died
Time Frame: From Day 1 to death from any cause, up to the study completion date (approximately 43 months)
Population: The efficacy-evaluable population included participants who received at least one dose of study drug. Data are reported for participants with events.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort IHC2+ | Cohort IHC3+
Number analyzed (Participants) | 29 | 20
percentage of participants | 79.3 | 80.0

3. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from first study drug administration to death from any cause.
Time Frame: From Day 1 to death from any cause, up to the study completion date (approximately 43 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort IHC2+ | Cohort IHC3+
Number analyzed (Participants) | 29 | 20
months | 12.2 [3.8 to 23.6] | 13.7 [4.1 to 33.0]

4. Secondary Outcome: Percentage of Participants With PFS Event of Disease Progression, as Per Investigator Assessment According to RECIST v. 1.1, or Death
Description: PFS is defined as the time from first study drug administration to first documented disease progression, based on investigator assessment using RECIST, v1.1, or death from any cause during the study, whichever occurs first. Disease progression is defined as: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study, including baseline; an absolute increase of at least 5 mm in the sum of diameters of target lesions; the appearance of one or more new lesions.
Time Frame: From Day 1 to PD or death from any cause, up to the study completion date (approximately 43 months)
Population: The efficacy-evaluable population included participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort IHC2+ | Cohort IHC3+
Number analyzed (Participants) | 29 | 20
percentage of participants | 100 | 95.0

5. Secondary Outcome: Progression-Free Survival (PFS) as Per Investigator Assessment According to RECIST v. 1.1
Description: as for outcome 4
Time Frame: From Day 1 to PD or death from any cause, up to the study completion date (approximately 43 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort IHC2+ | Cohort IHC3+
Number analyzed (Participants) | 29 | 20
months | 2.6 [1.4 to 2.8] | 2.7 [1.4 to 8.3]

6. Secondary Outcome: Percentage of Participants With DOR Event of Disease Progression, Assessed According to RECIST v1.1
Description: DOR is defined as the time from the initial documentation of response (CR or PR using RECIST, v1.1) to documented disease progression using RECIST v1.1 or death from any cause during the study. CR: disappearance of all target lesions; and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. Disease progression: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study, including baseline; an absolute increase of at least 5 mm in the sum of diameters of target lesions; the appearance of one or more new lesions.
Time Frame: From first documented objective response to PD or death from any cause, up to the study completion date (approximately 43 months)
Population: The efficacy-evaluable population included participants who received at least one dose of study drug. Data are reported for participants with response.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort IHC2+ | Cohort IHC3+
Number analyzed (Participants) | 0 | 4
percentage of participants |  | 75.0 [2.9 to 8.3]

7. Secondary Outcome: Duration of Objective Response (DOR) Assessed According to RECIST v1.1
Description: as for outcome 6
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort IHC2+ | Cohort IHC3+
Number analyzed (Participants) | 0 | 4
months |  | 7.3 [2.9 to NA] — The upper limit confidence interval was not calculable due to the low number of participants with events.

8. Secondary Outcome: Percentage of Participants With Clinical Benefit as Per Investigator Assessment According to RECIST, v1.1
Description: Clinical benefit is defined as having a CR or PR or stable disease (using RECIST, v1.1) at 6 months. Participants with no post-baseline response assessment are considered as experiencing no clinical benefit. CR: disappearance of all target lesions; and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. Stable disease: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression, taking as reference the smallest sum while in the study. Disease progression: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study, including baseline; an absolute increase of at least 5 mm in the sum of diameters of target lesions; the appearance of one or more new lesions.
Time Frame: From Day 1 to PD or death from any cause, up to the study completion date (approximately 43 months)
Population: The efficacy-evaluable population included participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort IHC2+ | Cohort IHC3+
Number analyzed (Participants) | 29 | 20
percentage of participants | 6.9 [0.85 to 22.77] | 30.0 [11.89 to 54.28]

9. Secondary Outcome: Percentage of Participants With Adverse Events (AEs) and Serious AEs (SAEs)
Description: An AE is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product, whether or not considered related to the study drug. A SAE is any experience that: results in death, is life-threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is medically significant.
Time Frame: From Day 1 to 30 days after last dose of study drug, up to the study completion date (approximately 43 months)
Population: The safety-evaluable population included participants who received at least one dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort IHC2+ | Cohort IHC3+
Number analyzed (Participants) | 29 | 20
percentage of participants
  AEs | 93.1 | 95.0
  SAEs | 17.2 | 25.0

10. Secondary Outcome: Maximum Observed Concentration (Cmax) for Trastuzumab Emtansine and Total Trastuzumab
Description: Cmax is the 0-21 day maximum observed concentration of a drug and was measured in blood serum.
Time Frame: Pre-dose (within 2 days) and 30 minutes (min) after end of infusion (infusion length= 100 min or less) on Day 1 of Cycles 1 and 3 (one cycle=21 days); at treatment discontinuation/early termination, up to primary analysis, approx. 22 months
Population: The pharmacokinetic (PK) population included participants who had received at least one dose of study treatment and had at least one serum or plasma concentration result available at clinical data cut-off. Data are reported for evaluable participants.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (ug/mL)
Groups:
- Pharmacokinetic (PK) Analysis Group: Participants with HER2 IHC2 or IHC3-positive (IHC 2+ or IHC 3+) locally advanced or metastatic NSCLC, who had received at least one prior platinum-based chemotherapy regimen, will receive trastuzumab emtansine.
Arm/Group | Pharmacokinetic (PK) Analysis Group
Number analyzed (Participants) | 44
micrograms per milliliter (ug/mL)
  Trastuzumab Emtansine | 78.7 (19.6)
  Total Trastuzumab | 79.9 (21.3)

11. Secondary Outcome: AUCinf for Trastuzumab Emtansine and Total Trastuzumab
Description: AUC (from zero to infinity) represents the total drug exposure over time in blood serum.
Time Frame: Pre-dose & 30 minutes (min) post-infusion (inf.) on Day (D) 1 of Cycles (C) 1 & 3; post- inf. on D 2, 3, 4 or 5, 8, & 15 of C 1, & pre- inf. on D1 of C2 & D1 of C 4 (C=21 D); at discontin./termination, up to primary analysis, approx. 22 months
Population: The pharmacokinetic (PK) population included participants who had received at least one dose of study treatment and had at least one serum or plasma concentration result available at clinical data cut-off. Data are reported for evaluable participants who consented to intense sampling.
Measure: Mean (Standard Deviation); unit: days times ug/mL (day* ug/mL)
Arm/Group | Pharmacokinetic (PK) Analysis Group
Number analyzed (Participants) | 4
days times ug/mL (day* ug/mL)
  Trastuzumab Emtansine | 324 (49.9)
  Total Trastuzumab | 436 (83.4)

12. Secondary Outcome: Elimination Half-Life (t1/2) for Trastuzumab Emtansine and Total Trastuzumab
Description: t1/2 is the time required for the drug serum concentration to be reduced to half.
Time Frame: Pre-dose & 30 minutes (min) post-infusion (inf.) on D 1 of C 1 & 3; post- inf. on D 2, 3, 4 or 5, 8, & 15 of C 1, & pre- inf. on D 1 of C 2 & D 1 of C 4 (C=21 days); at treatment discontin./early termination, up to primary analysis, approx. 22 months
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Pharmacokinetic (PK) Analysis Group
Number analyzed (Participants) | 4
days
  Trastuzumab Emtansine | 3.2 (0.51)
  Total Trastuzumab | 5.6 (1.14)

13. Secondary Outcome: Volume of Distribution (Vss) for Trastuzumab Emtansine and Total Trastuzumab
Description: Vss is the volume of distribution of study drug at steady state.
Time Frame: Pre-dose & 30 minutes (min) post-infusion (inf.) on D1 of C1 & 3; post- inf. on D2, 3, 4 or 5, 8, & 15 of C 1, & pre- inf. on D 1 of C 2 & D1 of C 4 (C=21 days); at treatment discontin/early termination, up to primary analysis, approx. 22 months
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: milliliters kilogram (mL/kg)
Arm/Group | Pharmacokinetic (PK) Analysis Group
Number analyzed (Participants) | 4
milliliters kilogram (mL/kg)
  Trastuzumab Emtansine | 51.1 (1.81)
  Total Trastuzumab | 60.7 (4.23)

14. Secondary Outcome: Clearance (CL) for Trastuzumab Emtansine and Total Trastuzumab
Description: CL is a measure of the body's elimination of a drug from blood serum over time.
Time Frame: Pre-dose & 30 minutes (min) post-infusion (inf.) on D 1 of C 1 & 3; post- inf. on D 2, 3, 4 or 5, 8, & 15 of C 1, & pre- inf. on D 1 of C 2 & D 1 of C 4 (C=21 days); at treatment discontin/early termination, up to primary analysis, approx. 22 months
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mL/day/kg
Arm/Group | Pharmacokinetic (PK) Analysis Group
Number analyzed (Participants) | 4
mL/day/kg
  Trastuzumab Emtansine | 11.35 (1.99)
  Total Trastuzumab | 8.54 (1.99)

15. Secondary Outcome: Maximum Observed Concentration (Cmax) for N2'- Deacetyl-N2'-(3-mercapto-1-oxopropyl)-Maytansine (DM1)
Description: Cmax is the maximum observed concentration of a drug and was measured in blood plasma.
Time Frame: Pre-dose (within 2 days) and 30 minutes (min) after end of infusion (infusion length= 100 min or less) on Day 1 of Cycle 1 (one cycle=21 days); at treatment discontinuation/early termination,up to primary analysis, approx. 22 months
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Pharmacokinetic (PK) Analysis Group
Number analyzed (Participants) | 34
nanograms per milliliter (ng/mL) | 4.3 (3.36)

16. Secondary Outcome: Percentage of Participants With Treatment-Emergent Anti-Drug Antibodies (ADAs)
Description: The presence of ADAs in blood serum is an indication of the body's immune response to a drug.
Time Frame: Pre-dose (within 2 days) on Day 1 of Cycles 1 and 3; at treatment discontinuation/early termination,up to primary analysis, approx. 22 months
Population: The pharmacokinetic (PK) population included participants who had received at least one dose of study treatment and had at least one serum or plasma concentration result available at clinical data cut-off. Data are reported for evaluable participants with post-dose sample available for ADA analysis.
Measure: Number; unit: percentage of participants
Groups:
- Anti-drug Antibody Analysis Group: Participants with HER2 IHC2 or IHC3-positive (IHC 2+ or IHC 3+) locally advanced or metastatic NSCLC, who had received at least one prior platinum-based chemotherapy regimen, will receive trastuzumab emtansine.
Arm/Group | Anti-drug Antibody Analysis Group
Number analyzed (Participants) | 39
percentage of participants | 0

ADVERSE EVENTS:
Time Frame: From baseline to study completion (approximately 43 months)
Arm/Group | Cohort IHC2+ | Cohort IHC3+
All-Cause Mortality (participants affected / at risk) | 23/29 | 16/20
Serious Adverse Events (participants affected / at risk) | 5/29 | 5/20
Other Adverse Events (participants affected / at risk) | 24/29 | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort IHC2+ (N=29) | Cohort IHC3+ (N=20)
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Seizure (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort IHC2+ (N=29) | Cohort IHC3+ (N=20)
Fatigue (General disorders) | 10 | 3
Asthenia (General disorders) | 5 | 4
Chills (General disorders) | 1 | 4
Pyrexia (General disorders) | 4 | 3
Chest pain (General disorders) | 0 | 2
Mucosal inflammation (General disorders) | 2 | 1
Malaise (General disorders) | 2 | 0
Oedema peripheral (General disorders) | 1 | 1
Influenza like illness (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Oedema (General disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 10 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 6 | 3
Vomiting (Gastrointestinal disorders) | 3 | 2
Dry mouth (Gastrointestinal disorders) | 4 | 0
Constipation (Gastrointestinal disorders) | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Mouth ulceration (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 3
Platelet count decreased (Investigations) | 2 | 2
Weight decreased (Investigations) | 3 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 4 | 1
Headache (Nervous system disorders) | 3 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 2
Paraesthesia (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 3
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 3 | 4
Skin Wound (Injury, poisoning and procedural complications) | 0 | 1
Respiratory tract infection (Infections and infestations) | 3 | 0
Urinary tract infection (Infections and infestations) | 1 | 2
Pneumonia (Infections and infestations) | 0 | 2
Paronychia (Infections and infestations) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 3
Anxiety (Psychiatric disorders) | 0 | 1
Depressive symptom (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 3
Sinus tachycardia (Cardiac disorders) | 1 | 1
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Poor venous access (Vascular disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 1
Mucosal Dryness (General disorders) | 0 | 1
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Iron Deficiency (Metabolism and nutrition disorders) | 2 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.